CLINICAL TRIAL: NCT00713193
Title: A Multi-Center, Randomized Study of Cyclosporine or Corticosteroids as an Adjunct to Plasma Exchange in the Initial Therapy of Thrombotic Thrombocytopenic Purpura (TTP)
Brief Title: Study of Cyclosporine or Corticosteroids as an Adjunct to Plasma Exchange in Thrombotic Thrombocytopenic Purpura (TTP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Spero Cataland, Professor of Internal Medicine, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007H0194; R01FD003932 (FDA)
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2023-04-28 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Thrombotic Thrombocytopenic Purpura
Keywords: Idiopathic TTP; Treatment; Exacerbation; Relapse; Plasma Exchange
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic; Recurrence | interventions — Cyclosporine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine and Plasma Exchange Arm (Experimental): Patients in this arm will receive cyclosporine (Neoral) at a dose of 2-3 mg/kg orally as an adjunct to plasma exchange.
  All patients initiated daily PEX (one plasma volume), using plasma as the replacement fluid. Patients randomized to the CSA arm received CSA at a dose of 2-3 mg/kg (rounded to the nearest 50 mg increment) divided into a twice daily dosing (Figure 1a). Patients randomized to CSA did not receive steroids, but were permitted to receive hydrocortisone as required for any hypersensitivity reactions to the infused plasma. Daily PEX was continued until a clinical response was achieved, then patients received PEX every other day for 2 additional procedures, with the first day that the platelet count and LDH were normal counting as the first of the 2 procedures.
  Interventions: Drug: Cyclosporine
- Prednisone and Plasma Exchange Arm (Active Comparator): Patients in this arm will receive prednisone at a dose of 1 mg/kg as an adjunct to plasma exchange.
  All patients initiated daily PEX (one plasma volume), using plasma as the replacement fluid. Patients randomized to the corticosteroid arm received prednisone at a dose of 1 mg/kg/d rounded to the nearest 20 mg increment. Daily PEX was continued until a clinical response was achieved, then patients received PEX every other day for 2 additional procedures, with the first day that the platelet count and LDH were normal counting as the first of the 2 procedures.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Cyclosporine — 2-3 mg/kg orally in a twice day divided dose for 6 months
  Other Names: Neoral
  Arms: Cyclosporine and Plasma Exchange Arm
Drug: Prednisone — 1 mg/kg orally, daily for at least 30 days, then tapered over 30 days after achieving remission.
  Other Names: Steroid arm
  Arms: Prednisone and Plasma Exchange Arm

SUMMARY:
This research involves the use of immune base therapy as an adjunct to plasma exchange, the present standard of care for thrombotic thrombocytopenic purpura (TTP). Funding source -FDA OOPD

DETAILED DESCRIPTION:
TTP is a rare blood disorder that causes blood clots to form in the small blood vessels throughout the body, including the kidneys, brain, abdomen, and the heart. Plasma exchange is the standard treatment for TTP. Plasma exchange is a treatment that removes the plasma (the liquid portion of the blood without any cells) from a patient and replaces it with plasma from a donor. With plasma exchange, 90% of patients achieve a remission of the disease. Unfortunately, up to one half of patient will relapse after the plasma exchange has stopped, leading to significant complications and added risks to the patient.

This study randomizes patients to receive either prednisone or cyclosporine as an adjunct to plasma exchange, with the cyclosporine arm being the experimental arm of the study. All patients will undergo plasma exchange but will be randomized to receive either prednisone or cyclosporine as an adjunct to plasma exchange. Previous studies suggested that cyclosporine was superior to prednisone as an adjunct to plasma exchange, and therefore this randomized study attempts to confirm the findings of two previous single institution studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of idiopathic TTP as defined by a microangiopathic hemolytic anemia and thrombocytopenia (<100 x 103)
* Additional components of the pentad (fever, renal and neurologic abnormalities) need not be present.
* Additional explanations for the microangiopathic changes including DIC and malignancy should be excluded.
* Patients with pregnancy associated TTP will be permitted on this therapeutic trial if the child is delivered prior to the initiation of therapy for TTP. However, female patients that are breastfeeding and are unwilling to discontinue breastfeeding at the time of enrollment will be excluded from this study
* Patients with a previous diagnosis of TTP are eligible to be enrolled provided they meet eligibility criteria and have not been treated for an TTP in the past 30 days
* Given the potential for nephrotoxicity with CSA, all patients must have a serum creatinine of < 2.5 mg/dl prior to enrollment

Exclusion Criteria:

* In light of concern for the prompt initiation of PE, all patients with suspected TTP may be enrolled on this trial. If it is subsequently found that the patient does not meet enrollment criteria, they will be removed and their spot replaced for study purposes. Patients removed from the study after enrollment will continue to be followed longitudinally for 6 months to be monitored for safety and will be included in the safety database.
* Patients with TTP clinically categorized as secondary to stem cell transplant and solid organ, bloody diarrhea associated, malignancy associated, and drug associated will not be enrolled on this therapeutic study.
* Incarcerated patients will be excluded from the study due to the inherent difficulties in maintaining close follow-up for study purposes in patients who are incarcerated.
* Any patients already being treated chronically with corticosteroids or cyclosporine and taking these at the time of their presentation will be excluded from this study.
* Female patients that are breastfeeding and are unwilling to discontinue breastfeeding at the time of enrollment will be excluded from this study
* Patients taking any medications contraindicated in combination with CSA that cannot be safely discontinued will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-11; Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spero R Cataland, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
data being evaluated and reviewed, manuscript in preparation for final report to FDA
Supporting Information: Study Protocol, CSR
Time Frame: Presently available to share
Access Criteria: Request needs to be made to investigators

REFERENCES:
- [Derived] Cataland SR, Kourlas PJ, Yang S, Geyer S, Witkoff L, Wu H, Masias C, George JN, Wu HM. Cyclosporine or steroids as an adjunct to plasma exchange in the treatment of immune-mediated thrombotic thrombocytopenic purpura. Blood Adv. 2017 Oct 23;1(23):2075-2082. doi: 10.1182/bloodadvances.2017009308. eCollection 2017 Oct 24. PMID 29296854

RESULTS

PARTICIPANT FLOW:
Groups:
- CSA Arm: Patients in this arm will receive cyclosporine (Neoral) at a dose of 2-3 mg/kg orally as an adjunct to plasma exchange.
  Cyclosporine: 2-3 mg/kg orally in a twice day divided dose for 6 months
  All patients initiated daily PEX (one plasma volume), using plasma as the replacement fluid. Patients randomized to the corticosteroid arm received prednisone at a dose of 1 mg/kg/d rounded to the nearest 20 mg increment. Patients randomized to the CSA arm received CSA at a dose of 2-3 mg/kg (rounded to the nearest 50 mg increment) divided into a twice daily dosing (Figure 1a). Patients randomized to CSA did not receive steroids, but were permitted to receive hydrocortisone as required for any hypersensitivity reactions to the infused plasma. Daily PEX was continued until a clinical response was achieved, then patients received PEX every other day for 2 additional procedures, with the first day that the platelet count and LDH were normal counting as the first of the 2 procedures.
- Prednisone Arm: Patients in this arm will receive prednisone at a dose of 1 mg/kg as an adjunct to plasma exchange.
  Prednisone: 1 mg/kg orally, daily for at least 30 days, then tapered over 30 days after achieving remission.
  All patients initiated daily PEX (one plasma volume), using plasma as the replacement fluid. Patients randomized to the corticosteroid arm received prednisone at a dose of 1 mg/kg/d rounded to the nearest 20 mg increment. Patients randomized to the CSA arm received CSA at a dose of 2-3 mg/kg (rounded to the nearest 50 mg increment) divided into a twice daily dosing (Figure 1a). Patients randomized to CSA did not receive steroids, but were permitted to receive hydrocortisone as required for any hypersensitivity reactions to the infused plasma. Daily PEX was continued until a clinical response was achieved, then patients received PEX every other day for 2 additional procedures
Period: Overall Study
Arm/Group | CSA Arm | Prednisone Arm
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CSA Arm: Patients in this arm will receive cyclosporine (Neoral) at a dose of 2-3 mg/kg orally as an adjunct to plasma exchange.
  At the time of diagnosis, patients will be started on daily cyclosporine (Neoral) therapy at a dose of 2-3 mg/kg/day (rounded to the nearest 50 mg increment) concurrent with daily plasma exchange. Doses will be administered in the capsule form. The total dose will be divided into twice daily dosing. For consistency and standardization of cyclosporine levels throughout the study, doses of Neoral (cyclosporine) should be given at 8 AM and 8 PM each day. Neoral (cyclosporine) should be taken on an empty stomach, and patients should not eat for at least 30 minutes after their dose of Neoral (cyclosporine). Cyclosporine will be continued for a total of six months of therapy and then discontinued.
- Prednisone Arm: Patients in this arm will receive prednisone at a dose of 1 mg/kg as an adjunct to plasma exchange.
  Prednisone: 1 mg/kg orally, daily for at least 30 days, then tapered over 30 days after achieving remission.
  At the time of diagnosis, patients will be started on daily prednisone therapy at a dose of 1 mg/kg/day (rounded off to the nearest 20 mg multiple) concurrently with daily PE. Patients unable to take oral corticosteroids will be switched to an equivalent intravenous corticosteroid until they are able to take oral medications. Patients may receive intravenous corticosteroids at any time to urgently treat reactions to the infused plasma and for prophylaxis against future reactions prior to the next TPE.
- Total: Total of all reporting groups
Arm/Group | CSA Arm | Prednisone Arm | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 40 [18 to 63] | 37 [22 to 63] | 37 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 14 | 16
  Male | 10 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 14 | 16
  White | 10 | 0 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Exacerbations in the CSA/PEX Arm Compared to the Steroids/PEX Arm
Description: Number of Participants with Exacerbations in the CSA/PEX Arm Compared to the Steroids/PEX Arm
Time Frame: From the start of treatment until 30 days after discharge from the last PEX procedure
Measure: Number; unit: participants
Groups:
- CSA Arm: Patients in this arm will receive cyclosporine (Neoral) at a dose of 2-3 mg/kg orally as an adjunct to plasma exchange.
  All patients initiated daily PEX (one plasma volume), using plasma as the replacement fluid. Patients randomized to the CSA arm received CSA at a dose of 2-3 mg/kg (rounded to the nearest 50 mg increment) divided into a twice daily dosing (Figure 1a). Patients randomized to CSA did not receive steroids, but were permitted to receive hydrocortisone as required for any hypersensitivity reactions to the infused plasma. Daily PEX was continued until a clinical response was achieved, then patients received PEX every other day for 2 additional procedures, with the first day that the platelet count and LDH were normal counting as the first of the 2 procedures.
  Cyclosporine: 2-3 mg/kg orally in a twice day divided dose for 6 months
- Prednisone Arm: Patients in this arm will receive prednisone at a dose of 1 mg/kg as an adjunct to plasma exchange.
  All patients initiated daily PEX (one plasma volume), using plasma as the replacement fluid. Patients randomized to the corticosteroid arm received prednisone at a dose of 1 mg/kg/d rounded to the nearest 20 mg increment. Daily PEX was continued until a clinical response was achieved, then patients received PEX every other day for 2 additional procedures, with the first day that the platelet count and LDH were normal counting as the first of the 2 procedures.
  Prednisone: 1 mg/kg orally, daily for at least 30 days, then tapered over 30 days after achieving remission.
Arm/Group | CSA Arm | Prednisone Arm
Number analyzed (Participants) | 12 | 14
participants | 3 | 1

2. Secondary Outcome: Time in Days to Achieve a Clinical Response, Comparing the CSA/PEX Arm to the Steroids/PEX Arm.
Description: Days to achieve a clinical response, defined as a normal platelet count (>150 x 109/L), normal LDH, and no new end organ injury.
Time Frame: Time to starting treatment until 6 months after the last PEX procedure
Measure: Median (Full Range); unit: Days
Arm/Group | CSA Arm | Prednisone Arm
Number analyzed (Participants) | 12 | 14
Days | 5 [4 to 19] | 5 [4 to 8]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected over the first 6 months
Arm/Group | CSA Arm | Prednisone Arm
All-Cause Mortality (participants affected / at risk) | 1/12 | 1/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-08-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT00713193/Prot_SAP_000.pdf